CLINICAL TRIAL: NCT03172520
Title: Use of Automatic Periodic Stimulation and Continuous EMG for Facial Nerve Monitoring During Parotidectomy
Brief Title: Automatic Periodic Stimulation and Continuous Electromyography (EMG) for Facial Nerve Monitoring During Parotidectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limitations in timing and personnel
Sponsor: Mayo Clinic (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Eric J. Moore, M.D., Professor of Otolaryngology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16-009380
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Parotid Gland Disorders
Keywords: Parotidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Facial Nerve Monitoring with APS electrode (Experimental): The investigators will use the Facial Nerve Monitor along with the automatic periodic stimulating(APS) electrode during parotidectomy surgery.
  Interventions: Device: APS electrode; Device: Facial Nerve Monitor

INTERVENTIONS:
Device: APS electrode — The APS electrode is an accessory intended for providing automatic periodic stimulation to nerves when used with the Medtronic Nerve Monitoring Systems.
  Other Names: automatic periodic stimulating (APS) Electrode Stimulator
Device: Facial Nerve Monitor — The facial nerve monitoring system records the number of stimulations of the facial nerve during the operation and this data is stored on the device until it is shut down after the surgery is complete.
  Other Names: NIM-Response 3.0

SUMMARY:
The purpose of this study is to document the safety of the Medtronic automatic periodic stimulating (APS) Electrode Stimulator during a parotidectomy and potentially prevent post-operative facial nerve weakness, which is a relatively common outcome after parotid surgery.

DETAILED DESCRIPTION:
This study will be conducted in two phases. In the first phase the investigators will use the same monitoring system currently used during parotidectomy and requires placement of the APS electrode as the only additional piece of equipment. During this phase, the investigators will record intraoperative EMG data generated by the monitoring system as well as document intra-operative maneuvers that precede adverse EMG events.

In the second phase of the study the investigators aim to allow the surgeon to alter his or her techniques, with the information provided by the APS electrode, to reverse adverse EMG changes.

ELIGIBILITY:
Inclusion Criteria:

* Parotidectomy: Planned parotid gland surgery (superficial or total parotidectomy)
* Benign or malignant disease

Exclusion Criteria:

* Current pregnancy
* Preoperative facial nerve dysfunction
* Revision surgery
* History of preoperative radiation to the surgical field
* Retrograde or extracapsular dissection
* Intentional nerve sacrifice (i.e., due to nerve involvement by tumor)
* Tumors with proximity to main trunk of facial nerve
* Inability to place electrode
* Presence of electrode alters surgical technique

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Moore, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Facial Nerve Monitoring With APS Electrode: The investigators will use the Facial Nerve Monitor along with the automatic periodic stimulating (APS) electrode during parotidectomy surgery.
  APS electrode: The APS electrode is an accessory intended for providing automatic periodic stimulation to nerves when used with the Medtronic Nerve Monitoring Systems.
  Facial Nerve Monitor: The facial nerve monitoring system records the number of stimulations of the facial nerve during the operation and this data is stored on the device until it is shut down after the surgery is complete.
Period: Overall Study
Arm/Group | Facial Nerve Monitoring With APS Electrode
Started | 10
Completed | 0
Not Completed | 10

BASELINE CHARACTERISTICS:
Groups:
- Facial Nerve Monitoring With APS Electrode: The investigators will use the Facial Nerve Monitor along with the APS electrode during parotidectomy surgery.
  APS electrode: The APS electrode is an accessory intended for providing automatic periodic stimulation to nerves when used with the Medtronic Nerve Monitoring Systems.
  Facial Nerve Monitor: The facial nerve monitoring system records the number of stimulations of the facial nerve during the operation and this data is stored on the device until it is shut down after the surgery is complete.
Arm/Group | Facial Nerve Monitoring With APS Electrode
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.67 (14.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Electromyography (EMG)
Description: EMG is an electrodiagnostic medicine technique for evaluating and recording the electrical activity produced by skeletal muscles.
Time Frame: baseline, approximately 3 hours
Population: Study terminated due to limitations in timing and personnel. Data was not collected
Arm/Group | Facial Nerve Monitoring With APS Electrode
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over a two day period.
Arm/Group | Facial Nerve Monitoring With APS Electrode
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT03172520/Prot_000.pdf